CLINICAL TRIAL: NCT03642327
Title: The Safe Environment for Every Kid (SEEK) Model: Dissemination and Implementation
Brief Title: SEEK: Dissemination and Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Chestnut Health Systems (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Howard Dubowitz, Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00078770
Record Dates: First submitted 2018-08-01; First posted 2018-08-22 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Child Maltreatment
Keywords: Child Abuse Prevention; Primary Care; Professional Education in Primary Care

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Independent online training (IND) (Active Comparator): IND refers to practitioners Independently doing the online training.
  Interventions: Other: Independent online training (IND)
- Maintenance of Certification (MOC) (Experimental): MOC involves a guided learning experience, approved by the American Board of Pediatrics and the American Board of Family Medicine for Maintenance of Certification credits. This involves a Quality Improvement project with 3 waves of data collection to assess and improve implementation while participating in 4 monthly webinars led by Dr. Dubowitz.
  Interventions: Behavioral: Experimental: Maintenance of Certification (MOC)

INTERVENTIONS:
Behavioral: Experimental: Maintenance of Certification (MOC) — MOC training will lead to more positive attitudes, comfort level and competence in addressing risk factors for Child Maltreatment.
  Arms: Maintenance of Certification (MOC)
Other: Independent online training (IND) — IND refers to practitioners Independently doing the online training.
  Arms: Independent online training (IND)

SUMMARY:
This study aims to understand what influences the adoption and implementation of an innovative approach to pediatric primary care by medical professionals and staff providing that care. The innovation concerns addressing common psychosocial problems such as parental depression and substance abuse. Different approaches to training medical professionals will be examined as well as the use of software versus traditional 'paper and pencil' to facilitate implementation.

DETAILED DESCRIPTION:
The proposed study, based on SEEK I and II findings is designed to study the effectiveness of technology driven training strategies to facilitate use of SEEK in helping prevent child maltreatment (CM) and its adoption and implementation in pediatric and family medicine settings. The implementation approach is anchored in four stages of the EPIS conceptual model: Exploration, adoption/Preparation, Implementation, and Sustainment. The strong evidence for SEEK's effectiveness has been underscored by its listing on the websites of the CDC, AHRQ, AAP, and by the California Clearinghouse for Evidence-Based Interventions in Child Welfare. Early adopters are increasingly implementing SEEK in primary care settings, including in Sweden. Four of the 5 healthcare systems in this proposal have implemented SEEK in some of their practices. However, practices within these systems operate independently of one another, and there should not be contamination among them. Each practice has its own lead physician, primary care providers (PCPs) and administrative staff and several have integrated behavioral health.

Design. The investigator selected a rigorous Hybrid Type III design which is an approach to examine implementation outcomes while also examining SEEK's effectiveness in preventing CM, measured by electron health record (EHR) indicators. Type III designs are facilitated by good EHR systems due to the low cost of data routinely gathered for clinical, services, and financial purposes. Five healthcare systems have committed to participating in the project, without committing individual practices and primary care providers (PCPs). Professionals, office staff and parents are nested within practices which are nested within the 5 participating healthcare systems. Practices will choose whether to participate, as will medical professionals within those practices. Participating practices will be randomized to one of the two training strategies for PCPs - Independent online training vs. a Maintenance of Certification (MOC) activity approved by the Boards of Pediatrics and of Family Physicians. Practices will be able to select the facilitation strategy (SEEKonline software or Traditional 'paper and pencil'). Participating professionals and staff within practices will need to adhere to the approach adopted by the practice. The design accounts for heterogeneity in geography, size of healthcare systems, type of primary care (pediatric and family medicine), and presence of integrated behavioral health. A small random sample of parents will be recruited from each practice.

For Aim 1, practices and PCPs will be randomized to one of the two training approaches. Using baseline and follow-up surveys, the investigators will assess the impact of each approach on PCPs' attitudes, knowledge, sense of competence, level of comfort and practice behavior with regard to addressing the targeted problems (e.g., parental depression).

Aim 2 focuses on the implementation of the SEEK model in pediatric and family medicine primary care practices. Practices will have the option of implementing the model using the SEEKonline software or the "traditional" paper and pencil approach. The evaluation involves measuring aspects of implementation such rates of adoption, fidelity to the model, and sustainment beyond the training. In addition, qualitative interviews will provide data regarding what facilitates or impedes optimal implementation.

For Aim 3, The investigators will assess the impact of the interventions on rates of child maltreatment (CM) based on ICD 10 diagnoses in EHRs. The investigators will include a cost-effectiveness analysis by estimating the costs associated with the different approaches to implementing SEEK.

ELIGIBILITY:
Inclusion Criteria:

* Practice not already implementing the SEEK model.
* The practice provides primary care to children.
* The practice agrees to participate in the study.
* PCPs, office staff and parents of children 0-5 years agree to participate.
* Able to comprehend basic English
* Access to a computer to complete online surveys.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dubowitz, MD, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubowitz H, Belanger R, Magder L, Palinkas LA, Kim H, Muralidharan V. Comparing 2 Training Modalities Supporting the Adoption of the Safe Environment for Every Kid Approach in Pediatric Primary Care. Acad Pediatr. 2025 Jan-Feb;25(1):102534. doi: 10.1016/j.acap.2024.07.001. Epub 2024 Jul 14. PMID 39004298
- [Background] Dubowitz H, Finkelhor D, Zolotor A, Kleven J, Davis N. Addressing Adverse Childhood Experiences in Primary Care: Challenges and Considerations. Pediatrics. 2022 Apr 1;149(4):e2021052641. doi: 10.1542/peds.2021-052641. PMID 35362065
- [Background] Dubowitz H, Saldana L, Magder LA, Palinkas LA, Landsverk JA, Belanger RL, Nwosu US. Protocol for comparing two training approaches for primary care professionals implementing the Safe Environment for Every Kid (SEEK) model. Implement Sci Commun. 2020 Sep 22;1:78. doi: 10.1186/s43058-020-00059-9. eCollection 2020. PMID 32974614
- [Background] Palinkas LA, Belanger R, Newton S, Saldana L, Landsverk J, Dubowitz H. Assessment of Adoption and Early Implementation Barriers and Facilitators of the Safe Environment for Every Kid (SEEK) Model. Acad Pediatr. 2023 Sep-Oct;23(7):1434-1445. doi: 10.1016/j.acap.2023.06.024. Epub 2023 Jun 22. PMID 37354951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric and family medicine practices across the U.S. were contacted from March 2019 to June 2022 through several avenues: American Academy of Pediatrics state chapters, collegial networks, healthcare system liaisons, and primary care networks. To be eligible, practices had to agree to randomization to either training modality and to introducing SEEK into their practice.
Pre-assignment Details: Of the 44 practices that expressed initial interest, 29 agreed to participation. Four withdrew prior to randomization, so 25 practices were randomized to IND (13) or MOC (12), stratified by practice type (family medicine/pediatrics) and resident training site (yes/no). 6 additional practices withdrew early on. Reasons included feeling already overwhelmed, compounded by the pandemic; the sole family medicine practice cited plans for universal screening within their healthcare system.
Units Other Than Participants: Practices randomly assigned to IND
Groups:
- Independent Online Training (IND): IND refers to practices where all its primary care professionals (PCPs)were randomly assigned to Independently doing the online training.
- Maintenance of Certification (MOC): MOC refers to the practices where all its PCPs were randomly assigned to do the Maintenance of Certification (MOC) - 4 training, approved by the American Board of Pediatrics.
Period: Overall Study
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Started | 148; 13 Practices randomly assigned to IND (Participants were in these categories: 1) primary care professionals (PCPs), 2) Behavioral health professionals (BHPs), 3) admin/nursing staff and 4) parents. Some analyses were at a practice level. No patients or children were recruited.) | 212; 12 Practices randomly assigned to IND
PCPs | 90; 13 Practices randomly assigned to IND | 120; 12 Practices randomly assigned to IND
Behavioral Health | 2; 13 Practices randomly assigned to IND | 9; 12 Practices randomly assigned to IND
Admin/Nursing | 11; 13 Practices randomly assigned to IND | 20; 12 Practices randomly assigned to IND
Parents | 45; 13 Practices randomly assigned to IND | 63; 12 Practices randomly assigned to IND
Completed (3 IND and 3 MOC practices withdrew participation due to the Covid 19 pandemic.) | 67; 10 Practices randomly assigned to IND | 93; 9 Practices randomly assigned to IND
Not Completed | 81; 3 Practices randomly assigned to IND | 119; 3 Practices randomly assigned to IND

BASELINE CHARACTERISTICS:
Population: Baseline demographic data was only collected on the PCPs.
Units Other Than Participants: Practices
Groups:
- Independent Online Training (IND): IND refers to practitioners independently doing the online training per practice assignment.
  We did not conduct separate analyses on the other subsamples: practice leaders, behavioral health professionals, admin/nursing and parents. Particularly in the 1st three groups the n was too low.
- Maintenance of Certification (MOC): MOC refers to practitioners trained via the SEEK MOC-4 Activity per practice assignment. involves a guided learning experience, approved by the American Board of Pediatrics and the American Board of Family Medicine for Maintenance of Certification credits. This involves a Quality Improvement project with 3 waves of data collection to assess and improve implementation while participating in 4 monthly webinars led by Dr. Dubowitz.
  We did not conduct separate analyses on the other subsamples: practice leaders, behavioral health professionals, admin/nursing and parents. Particularly in the 1st three groups the n was too low.
- Total: Total of all reporting groups
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC) | Total
Number analyzed (Participants) | 90 | 120 | 210
Number analyzed (Practices) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 120 | 210
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The difference between the numbers is that we only had adequate data on the analysis sample.
  Participants
    Sex: Female | 71 | 95 | 166
    Sex: Male | 19 | 25 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 10 | 14
  Not Hispanic or Latino | 84 | 108 | 192
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 23 | 23 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 55 | 80 | 135
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Count of Participants; unit: Participants] — Practices across the U.S. were recruited.
  Participants
    United States | 90 | 120 | 210

OUTCOME MEASURES:

1. Primary Outcome: Stages of SEEK Implementation Completion (SIC) - Startup (at a Practice Level)
Description: The SIC is an assessment tool with 8 stages extending from Engagement to achievement of Competency. Each stage maps onto 3 phases of implementation (Pre-Implementation, Implementation and Sustainment).
  Startup reflects whether the practice implemented SEEK - Yes/No. Yes = practice started implemented SEEK. Practices that did start are reported.
Time Frame: up to 30 months
Measure: Number; unit: practices
Units Other Than Participants: practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (practices) | 13 | 12
practices | 10 | 9

2. Primary Outcome: Stages of Implementation Completion (SIC) - as Assessed by the Safe Environment for Every Kid (SEEK) Fidelity Score (at a Practice Level)
Description: The SIC is an assessment tool with 8 stages extending from Engagement to achievement of Fidelity. Each stage maps onto 3 phases of implementation (Pre-Implementation, Implementation and Sustainment).
  Competence/Fidelity score reflects the extent to which a practice implemented the intervention as intended. Score range: 0-100; higher is better fidelity to the intervention as planned.
Time Frame: up to 30 months
Population: The n is different because 6 practices dropped out early on and were not included in the analyses.
  3 dropped out from each arm.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 10 | 9
Score on a scale | 90.4 (6.9) | 91.0 (6.5)

3. Primary Outcome: Stages of SEEK Implementation Completion (SIC) - Sustainability
Description: The SIC is an assessment tool with 8 stages extending from Engagement to achievement of Competency. Each stage maps onto 3 phases of implementation (Pre-Implementation, Implementation and Sustainability).
  Sustainability was determined if the practice was implementing SEEK 24 months after initiation and doing so with fidelity.
  Reporting the number of practices that achieved sustainability.
Time Frame: up to 30 months
Population: as for outcome 2
Measure: Number; unit: practices
Units Other Than Participants: practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (practices) | 10 | 9
practices | 6 | 8

4. Secondary Outcome: Overall Rates of Children With Possible Abuse and Neglect.
Description: International Classification of Diseases - 10 (ICD-10) codes related to possible child maltreatment (CM or child abuse and neglect) are readily accessible through EHRs. De-identified aggregate data were gathered towards the end of the study for all children in the practice 0-66 months of age.
Time Frame: 2 years prior to implementing SEEK, 2 years after implementing SEEK., 48 months total.
Population: Electronic Health Record (EHR) data were collected from 14 of the participating practices.
Measure: Number; unit: percentage of patients
Units Other Than Participants: Practices
Groups:
- Independent Online Training (IND): IND refers to practices where the clinicians were assigned to the IND training. n = 13
- Maintenance of Certification (MOC): MOC refers to practices where clinicians were assigned to the MOC training. (n = 12).
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 6 | 8
percentage of patients
  Pre-SEEK | 4.1 | 8.2
  Post-SEEK | 4.3 | 9.3

5. Secondary Outcome: Rates of Children With Possible Neglect.
Description: ICD-10 codes related to possible maltreatment (child abuse and neglect) are readily accessible through EHRs. De-identified aggregate data were gathered towards the end of the study for all children in the practice 0-66 months of age.
Time Frame: 2 years prior to implementing SEEK, 2 years after implementing SEEK., 48 months total.
Population: EHR data were collected from 14 of the participating practices.
Measure: Number; unit: percentage of patients
Units Other Than Participants: Practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 6 | 8
percentage of patients
  Pre-SEEK | 3.3 | 7.0
  Post-SEEK | 3.6 | 8.3

6. Secondary Outcome: Rates of Children With Non-adherence to Medical Care
Description: as for outcome 5
Time Frame: 2 years prior to implementing SEEK, 2 years after implementing SEEK., 48 months total.
Population: EHR data were collected from 14 of the participating practices.
Measure: Number; unit: percentage of patients
Units Other Than Participants: Practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 6 | 8
percentage of patients
  Pre-SEEK | 0.02 | 0.1
  Post-SEEK | 0.01 | 0.05

7. Secondary Outcome: Rates of Under Immunized Children
Description: as for outcome 5
Time Frame: 2 years prior to implementing SEEK, 2 years after implementing SEEK., 48 months total.
Population: EHR data were collected from 14 of the participating practices.
Measure: Number; unit: percentage of patients
Units Other Than Participants: Practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 6 | 8
percentage of patients
  Pre-SEEK | 0.009 | 0.02
  Post-SEEK | 0.01 | 0.018

8. Secondary Outcome: Rates of Children With Possible Abuse.
Description: as for outcome 5
Time Frame: 2 years prior to implementing SEEK, 2 years after implementing SEEK., 48 months total.
Population: EHR data were collected from 14 of the participating practices.
Measure: Number; unit: percentage of patients
Units Other Than Participants: Practices
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 148 | 212
Number analyzed (Practices) | 6 | 8
percentage of patients
  Pre-SEEK | 0.8 | 1.3
  Post-SEEK | 0.7 | 1.2

9. Secondary Outcome: The Safe Environment for Every Kid (SEEK) PCP Questionnaire (PCPQ) - Addressing Depression Subscale
Description: The PCPQ, used in both SEEK RCTs has 5 vignettes, with 7-12 statements assessing PCPs' thinking and practice with regard to addressing the targeted CM risk factors. Items were grouped conceptually into 6 topical scales (e.g., Substance Abuse) and 5 cross-cutting themes (e.g., Perceived Competence).
  The mean subscale scores ranged from 0-3. Higher scores reflect PCPs more optimal capability to address the problem.
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Independent Online Training (IND): IND refers to practitioners Independently doing the online training. n = 90.
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.12 (0.36) | 2.08 (0.41)

10. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Addressing Food Insecurity
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.19 (0.35) | 2.09 (0.41)

11. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Addressing Major Stress
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 1.93 (0.35) | 1.98 (0.39)

12. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Addressing Intimate Partner Violence
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.14 (0.40) | 2.02 (0.35)

13. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Addressing Harsh Punishment
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.16 (0.35) | 2.26 (0.31)

14. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Addressing Substance Abuse
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 1.98 (0.34) | 1.94 (0.31)

15. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Attitudes Regarding Addressing Health-related Social Needs
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.33 (0.32) | 2.26 (0.30)

16. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Comfort Level Regarding Addressing Health-related Social Needs
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.02 (0.40) | 1.99 (0.43)

17. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Perceived Competence Regarding Addressing Health-related Social Needs
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 1.78 (0.41) | 1.73 (0.43)

18. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Knowledge Regarding Addressing Health-related Social Needs
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.26 (0.28) | 2.21 (0.27)

19. Secondary Outcome: SEEK PCP Questionnaire (PCPQ) - Practice Behavior Regarding Addressing Health-related Social Needs
Description: as for outcome 9
Time Frame: 30 months
Population: The analysis is based on PCPs with data collected between 8 - 24 months after startup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 70 | 95
units on a scale | 2.07 (0.39) | 2.04 (0.40)

20. Secondary Outcome: SEEK Parent View of Relationship With Child's PCP Subscale - Adapted From the Patient-Doctor Interaction Scale
Description: Parents rate their child's PCP on this measure adapted for pediatric practice from the Patient-Doctor Interaction Scale. The Likert scale included 8 questions; the response set was from 1 (no) to 4 (always).
  Subscale mean scores range from 1 - 4; higher scores indicate greater satisfaction.
  The mean of the Likert subscale response is reported.
Time Frame: 24 months
Population: Represents all the data collected from parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Independent Online Training (IND): IND refers to parents in practices where clinicians completed the training independently online. n = 45
- Maintenance of Certification (MOC): MOC refers to parents in practices where clinicians completed training by a MOC-4 SEEK Activity approved by the American Board of Pediatrics. n = 63.
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 45 | 63
score on a scale | 3.53 (0.50) | 3.48 (0.44)

21. Secondary Outcome: SEEK Parent View of the Attentiveness of the Child's PCP Subscale - Adapted From the Patient-Doctor Interaction Scale
Description: as for outcome 20
Time Frame: 24 months
Population: Represents all the data collected from parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 45 | 63
score on a scale | 3.67 (0.38) | 3.62 (0.44)

22. Secondary Outcome: SEEK Parent View of the Comprehensiveness of the Child's PCP Subscale - Adapted From the Patient-Doctor Interaction Scale
Description: as for outcome 20
Time Frame: 24 months
Population: Represents all the data collected from parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 45 | 63
score on a scale | 3.08 (0.56) | 2.92 (0.56)

23. Secondary Outcome: SEEK Parent View of the Communication Skills of the Child's PCP Subscale - Adapted From the Patient-Doctor Interaction Scale
Description: as for outcome 20
Time Frame: 24 months
Population: Represents all the data collected from parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
Number analyzed (Participants) | 45 | 63
score on a scale | 3.61 (0.41) | 3.51 (0.43)

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Arm/Group | Independent Online Training (IND) | Maintenance of Certification (MOC)
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/212
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/212
Other Adverse Events (participants affected / at risk) | 0/148 | 0/212

LIMITATIONS AND CAVEATS:
The Covid pandemic affected practices and personnel and consequently the study. The sample is relatively small. ICD-codes from EHR data are a limited proxy for possible child abuse and neglect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT03642327/Prot_SAP_000.pdf